CLINICAL TRIAL: NCT02371551
Title: Evaluation of Complex Renal Cystic Lesions With Contrast Enhanced Ultrasound (CEUS) and Functional MRI Versus the Gold Standard: Computer Tomography (CT)
Brief Title: Evaluation of Complex Renal Cyst With CEUS/Functional MRI Versus CT
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 84/14
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Cystic Renal Diseases; Kidney Neoplasms
Keywords: Diffusion Magnetic Resonance Imaging; Medical Sonography; Computed Tomography, X-Ray
MeSH Terms: conditions — Kidney Diseases, Cystic; Kidney Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All patients
  Interventions: Other: Blood/urine sampling; Other: Conventional routine CT examination; Other: Contrast-enhanced renal ultrasonography (CEUS); Other: Functional MRI

INTERVENTIONS:
Other: Blood/urine sampling — Routine chemistry profile
Other: Conventional routine CT examination — Standard diagnostic examination
Other: Contrast-enhanced renal ultrasonography (CEUS) — Study-specific diagnostic examination
Other: Functional MRI — Study-specific diagnostic examination

SUMMARY:
The primary concern in complex renal cysts (CRC) with malignant potential is the accurate diagnosis and characterization. Patients with CRC have to undergo frequent imaging surveillance (every 6-12 Mo), in which the progression suggests a neoplastic process. The gold standard for establishing diagnosis and necessity for surgical intervention (i.e. partial nephrectomy) is conventional computer tomography (CT) imaging. Its main drawback is the radiation dose to the body and intravenous contrast media administration, which has a risk of nephrotoxicity.

Magnetic resonance imaging (MRI) with special functional sequences (fMRI) and contrast-enhanced ultrasonography (CEUS) allow measuring tissue blood flow and perfusion characteristics without ionizing radiation or nephrotoxic contrast media. To compare the diagnostic accuracy, sensitivity and specificity of CEUS/functional MRI versus the gold standard CT, 60 patients with CRC will be evaluated using all these 3 modalities. The main hypothesis is that fMRI and CEUS have equal accuracy with CT regarding diagnosis and classification of CRC lesions.

DETAILED DESCRIPTION:
Background

Renal cysts occur in a variety of diseases but also in normal kidneys (i.e. simple cysts). Diagnostic imaging plays a central role in the diagnosis of renal cysts and lesions. Most patients are diagnosed after undergoing imaging (computed tomography [CT], magnetic resonance imaging [MRI], ultrasound [US]) for an unrelated reason and their increasing incidental finding during the last decade parallels the growing use of imaging procedures.

Simple renal cysts are commonly observed in normal kidneys and are of limited clinical relevance. The primary clinical concern is the accurate evaluation of complex renal cysts (CRC) that have a malignant potential. Based upon the initial radiographic evaluation, further studies may be required, and some complex lesions may require surgical excision for exact diagnosis, based on growth during follow up.

The gold standard for the diagnosis of CRC is conventional CT imaging. Its main drawback is the radiation dose to the body and intravenous contrast media administration, which has a risk of nephrotoxicity. In order to accurate classify and manage these lesions, the Bosniak renal cyst classification system was created. Based upon morphologic and enhancement characteristics of the CT scan, cystic renal masses are placed in one of five categories (I, II, IIF, III, IV).

Although not yet validated for reader agreement or generalizability, the Bosniak renal cyst classification system has been widely accepted by urologists and radiologists as the best way to assess and follow these CRC lesions. While the Bosniak classification is based on CT findings, the same approach is applicable as a useful predefined framework for the evaluation of CRC with other radiographic modalities i.e. with MRI and conventional or contrast-enhanced ultrasound. The ability to differentiate between those that are benign versus malignant (surgical versus nonsurgical masses) still represents a major challenge.

Magnetic resonance imaging (MRI) has gained immense popularity over the last decades as it allows generation of very high-resolution images, including 3D reconstructions, without ionizing radiation. Functional MRI can be performed with or without injection of contrast, thus avoiding the risk of nephrogenic systemic sclerosis in patients with chronic kidney disease (CKD). Diffusion weighted imaging (DW-MRI), blood-oxygen-level-dependent (BOLD) MRI and arterial spin labeling (ASL) sequences are functional sequences which can be performed without injection of contrast.

The recent development and availability of a contrast-enhanced ultrasonography (CEUS) using microbubbles has further improved sensitivity and diagnostic confidence with respect to conventional and colour-Doppler US. They allow vascular bed opacification and have opened the way to detecting the microcirculation. CEUS was able to detect changes in human renal cortical microcirculation. Thus it seems to be a feasible technique to evaluate (i.e. perfusion pattern of the cyst wall or perfusion of the septa) CRC using the Bosniak classification system.

Ideally, the method for the evaluation of CRC should be safe, non-invasive, and accurate. Abdominal CT scanning delivers significant ionizing radiation, which may be a consideration for younger patients (age <35 years), utilizes contrast media with a considerable nephrotoxicity and risk of an allergic reaction. No prospective study comparing CT with CEUS or functional MRI for the evaluation of CRC has been conducted.

Objective

The primary aim of this study is to evaluate the diagnostic accuracy, sensitivity and specificity of CEUS/fMRI and compare it with abdominal CT the current gold standard diagnostic modality.

Methods

Prospective, single center, observational setting. Patients with CRC who fulfill the inclusion criteria will be further evaluated after written informed consent. Kidney function and the CRC progression will be followed according to the current medical standards. If a significant change in cystic lesions is observed, further evaluation and surgical intervention, if indicated, will be initiated by the primary physician in charge. Testing will be performed upon study entry and after 12 months according to the following schedule:

* Blood-sampling
* CT
* fMRI
* renal CEUS
* chart review Two study physicians independently will review the CEUS and functional MRI images of the patients. The reviewers will be aware of study design but will be blinded to the clinical information of the CT findings. The scoring system for image interpretation will be based on the Bosniak cyst classification.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Written informed consent
* A complicated renal cyst (Bosniak category > II cyst or hemorrhagic cyst) or lesion > 1 cm im max. transverse diameter who will undergo standard renal CT imaging
* Stable renal function (GFR> 30 ml/min/1.73 m2)

Exclusion Criteria

* Pregnancy
* History of allergic reaction to contrast agents
* Refusal to adhere to follow-up
* Recent pyelonephritis
* Acute kidney injury (AKI stage ≥ 1)
* Other individuals especially in need of protection (according to the Swiss Academy of Medical Sciences)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were referred to the outpatient clinic of the Department of Nephrology or to the Department of Urology, Bern University Hospital for the clarification of a complex renal cyst/lesion and already underwent or will undergo a standard CT examination or patient who where accidentally diagnosed with a complicated renal cyst/lesion from the Department of Nephrology, Urology or Radiology (with CT imaging)
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
CRC classification according to CT-finding based on Bosniak criteria or until surgical intervention | 1 year

SECONDARY OUTCOMES:
Diagnostic accuracy of CEUS and fMRI based on the progression of CRC according to CT-finding and Bosniak classification throughout visit 1-2 | 1 year
Diagnostic accuracy of CEUS and fMRI based on surgical extraction and histopathological evaluation of the resected mass | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Spyridon Arampatzis, MD, Principal Investigator — Dep. of Nephrology, Hypertension and Clinical Pharmacology, Bern University Hospital
Locations (1):
- Dep. of Nephrology, Hypertension and Clinical Pharmacology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Bosniak MA. Diagnosis and management of patients with complicated cystic lesions of the kidney. AJR Am J Roentgenol. 1997 Sep;169(3):819-21. doi: 10.2214/ajr.169.3.9275903. No abstract available.
- [Background] Curry NS, Cochran ST, Bissada NK. Cystic renal masses: accurate Bosniak classification requires adequate renal CT. AJR Am J Roentgenol. 2000 Aug;175(2):339-42. doi: 10.2214/ajr.175.2.1750339. PMID 10915671
- [Background] Balci NC, Semelka RC, Patt RH, Dubois D, Freeman JA, Gomez-Caminero A, Woosley JT. Complex renal cysts: findings on MR imaging. AJR Am J Roentgenol. 1999 Jun;172(6):1495-500. doi: 10.2214/ajr.172.6.10350279.
- [Background] Nicolau C, Bunesch L, Sebastia C. Renal complex cysts in adults: contrast-enhanced ultrasound. Abdom Imaging. 2011 Dec;36(6):742-52. doi: 10.1007/s00261-011-9727-8. PMID 21461960
- [Background] Schneider AG, Hofmann L, Wuerzner G, Glatz N, Maillard M, Meuwly JY, Eggimann P, Burnier M, Vogt B. Renal perfusion evaluation with contrast-enhanced ultrasonography. Nephrol Dial Transplant. 2012 Feb;27(2):674-81. doi: 10.1093/ndt/gfr345. Epub 2011 Jun 20. PMID 21690200